CLINICAL TRIAL: NCT04726059
Title: Motor and Autonomic Concomitant Health Improvements With Neuromodulation and Exercise (MACHINE) Training: A Randomized Controlled Trial in Individuals With SCI
Brief Title: Motor & Autonomic Concomitant Health Improvements With Neuromodulation & Exercise Training: An SCI RCT
Acronym: MACHINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Praxis Spinal Cord Institute (Other)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-01307
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder; Neurogenic Bowel
Keywords: Activity-based Therapy; Spinal Cord Stimulation; Transcutaneous Spinal Cord Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Neurogenic Bowel

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either an ABT+TSCS or ABT+SHAM arm. Participants who are assigned to ABT+SHAM will have the opportunity to complete an ABT+TSCS open-label follow-up.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABT+SHAM (Sham Comparator): The SHAM is low-intensity, ineffective stimulation delivered at the same anatomical location as TSCS.
  Interventions: Device: SHAM (low-intensity) Transcutaneous Spinal Cord Stimulation; Device: Activity-Based Therapy
- ABT+TSCS (Experimental): Therapeutic TSCS will be delivered during ABT using an isolated bipolar constant current stimulator. Continuous TSCS applied over the T11-T12 spinous processes at 5-40 Hz has been shown to induce stepping movements in participants with their legs in a gravity-independent position.
  Interventions: Device: Transcutaneous Spinal Cord Stimulation; Device: Activity-Based Therapy

INTERVENTIONS:
Device: Transcutaneous Spinal Cord Stimulation — Therapeutic TSCS will be delivered during ABT using a non-invasive central nervous system stimulator (TESCoN, SpineX Inc., CA, USA). Stimulation will involve charge balanced monophasic rectangular waveforms with 1.0-ms pulses, administered at 30 Hz, with a carrier frequency of 10 kHz and a current ranging from 10 to 130 mA.
  Arms: ABT+TSCS
Device: SHAM (low-intensity) Transcutaneous Spinal Cord Stimulation — Ineffective stimulation will be administered at the same anatomical location as therapeutic TSCS.
  Arms: ABT+SHAM
Device: Activity-Based Therapy — Using BWSTT, all participants (both arms) will train 3 times per week for 12 weeks with a target to reach 45 minutes of gait training in each session.
  For gait training, the level of body weight support and speed of walking will be adjusted to allow the person to bear as much weight as possible while maintaining proper stance limb kinematics.

SUMMARY:
Spinal cord injury (SCI) disrupts many aspects of life, including the loss of volitional movement and involuntary control of bodily functions; both crucial functional recovery priorities for this population. Mobility impairments and secondary complications limit an individual's ability to exercise, a behavior known to have wide-ranging functional and health benefits. This trial will investigate whether activity-based therapy (ABT), using body-weight-supported treadmill training (BWSTT), can change the strength of signals from the brain that control volitional movement, leading to improvements in seated balance as well as other important involuntary bodily (i.e. cardiovascular, urinary tract, bowel and sexual) functions. The investigators aim to determine whether these improvements can be augmented with the addition of non-invasive transcutaneous spinal cord stimulation (TSCS). This therapy has been shown to re-awaken dormant spinal circuits. In this randomized controlled trial, TSCS with ABT, using BWSTT (three sessions/week for twelve weeks), will be compared to ABT+SHAM in individuals with chronic motor-complete spinal cord injury (SCI). Those in the ABT+SHAM group will be given the option to complete an ABT+TSCS open-label follow-up. Before and after training, the following outcomes will be assessed by validated methods: corticospinal excitability, motor function, and seated balance (Hypothesis 1 - Motor Function); severity and frequency of blood pressure instability, urinary tract, bowel, and sexual dysfunctions (Hypothesis 2 - Autonomic Functions); and general health (Hypothesis 3 - Quality of Life). This collaborative project is between consumers with SCI and clinicians/scientists with expertise in SCI care (kinesiologists, physiotherapists, physiatrists, sexual health clinicians). Compared to ABT alone, the investigators anticipate that ABT+TSCS will result in superior improvements in motor and autonomic functions in individuals with SCI.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a severe disorder resulting in not only in motor deficits (i.e. paralysis) but also a myriad of autonomic dysfunctions (i.e. urinary tract/bowel/sexual impairments and blood pressure instability). The restoration of motor as well as autonomic functions remains among the top priorities for individuals with SCI. Individuals with SCI develop cardiovascular (CV) disease at a younger age and at greater rates than individuals without injury. Both low levels of physical activity and profound blood pressure (BP) instability, commonly experienced by individuals with injuries at or above the sixth thoracic level, likely explains the heightened risk.

Neurogenic lower urinary tract (LUT) dysfunction impacts over 90% of individuals with SCI. This dysfunction leads to vesico-ureteral-renal reflux, urinary tract infections, bladder stone formation, and impaired renal function - ultimately leading to significant disease burden and poorer health-related quality of life. Bowel function is also significantly compromised after SCI, presenting as constipation, impaired colonic motility and loss of volitional control resulting in episodes of fecal incontinence - predisposing an individual to increased risk of long-term complications. Over 60% report that bowel dysfunction adversely impacts quality of life. Lastly, severe impairments in sexual function following SCI include erectile dysfunction, ejaculatory disorders/ anejaculation in men and reduced vaginal lubrication in women, with both sexes experiencing orgasmic difficulties or anorgasmia as well as alterations in sexual drive and sexual satisfaction.

Activity-based therapy (ABT) is a common and an effective means to improve walking function post-injury and can facilitate general health maintenance; this includes an enhancement of neural BP control, as well as bladder, bowel, and sexual functions.

Neuromodulation, potentially activating isolated spinal cord neuronal circuitry, has received significant recognition in recent years as a promising approach to target various neurological dysfunctions. The immense therapeutic potential of epidural spinal cord stimulation demonstrates mitigation of spasticity in individuals with motor-incomplete injuries. Moreover, this stimulation improved ability to generate rhythmic, locomotor-like limb movements, and restored voluntary control of functional movements in individuals with motor-complete injuries. Our past exciting and ground-breaking pilot work highlights the capacity for TSCS to modulate spinal circuits (An Autonomic Neuroprosthesis: Noninvasive Electrical Spinal Cord Stimulation Restores Autonomic Cardiovascular Function in Individuals with Spinal Cord Injury. J Neurotrauma. 2018;35(3):446- 451. doi:10.1089/neu.2017.5082). To administer TSCS, small adhesive electrodes are placed on the skin around the spinal cord and hips. The electrodes are connected to a machine that generates a small electric current. After turning the machine on, the participant may feel a small electric current under the electrodes, though it should not elicit any pain.

Despite literature supporting the benefits of TSCS and ABT, the effects of pairing TSCS with ABT is largely unknown. These therapies are adaptable, non-invasive, and relatively affordable, with the potential to simultaneously benefit both motor and autonomic functions. Randomized controlled trials are needed to better validate these interventions for clinical settings.

Project Rationale:

Motor paralysis and autonomic dysfunctions have been identified as a major priority for recovery by individuals with SCI. Addressing these dysfunctions may ultimately translate to improved health-related quality of life (HRQOL). The use of ABT with non-invasive and adaptable TSCS has the potential to reduce CV disease risk factors and other autonomic dysfunctions in this at-risk population.

ELIGIBILITY:
INCLUSION CRITERIA

A participant must meet all of the following criteria in order to be eligible for inclusion:

* Resident of British Columbia, Canada with active provincial medical services plan
* Male or female, 18-60 years of age
* Chronic traumatic SCI (non-progressive, with complete motor paralysis) at or above the T6 spinal segment
* At least 1-year post injury, at least 6 months from any spinal surgery
* American Spinal Injury Association Impairment Scale (AIS) A, B
* Able to tolerate an upright posture for 30 minutes (with or without breaks)
* Willing and able to comply with all clinic visits and study-related procedures
* Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator)
* No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or active infection that may interfere with testing activities
* Stable management of spinal cord related clinical issues (i.e., spasticity management)
* Women of childbearing potential must not be intending to become pregnant, currently pregnant, or lactating. The following conditions apply:

  1. Women of childbearing potential must have a confirmed negative pregnancy test prior to the baseline visit. During the trial, all women of childbearing potential will undergo urine pregnancy tests at their monthly clinic visits as outlined in the schedule of events
  2. Women of childbearing potential must agree to use adequate contraception during the period of the trial and for at least 28 days after completion of treatment. Effective contraception includes abstinence
* Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment
* Medication dosage must be stable for period of 4 weeks prior to participation
* Must provide informed consent

EXCLUSION CRITERIA

A participant who meets any of the following criteria will be ineligible to participate:

* Ventilator dependent
* Clinically significant, unmanaged, depression (PHQ-9 above 15) or ongoing drug abuse
* Use of any medication or treatment that in the opinion of the investigator indicates that it is not in the best interest of the participant to participate in this study
* Intrathecal baclofen pump
* Oral baclofen dose or other anti-spasticity medications greater than 30mg per day
* Cardiovascular, respiratory, bladder, or renal disease unrelated to SCI or presence of hydronephrosis or presence of obstructive renal stones
* Presence of severe acute medical issue that in the investigator's judgement would adversely affect the participant's participation in the study. Examples include, but are not limited to acute urinary tract infections, active heterotopic ossification, newly changed antidepressant medications [tricyclics], debilitating muscle pain, pressure sores, or unstable diabetes
* Any implanted metal (other than dental implants) in the skull or presence of pacemakers, stimulators, or medication pumps in the trunk
* History of osteoporosis, low bone mineral density, or fragility fractures in the lower limbs
* History of seizures/epilepsy or recurring headaches
* Participant has swollen, infected, and inflamed areas or open wounds on the area of stimulation
* Severe anemia (Hgb<8 g/dl) or hypovolemia as measured by hematocrit via blood test in the last six months
* Participant is a member of the investigational team or his /her immediate family
* Participant has undergone electrode implantation surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in attempted voluntary motor activation (supine) | Weeks 2 and 14
  While lying in the supine position, the following voluntary motor contractions will be attempted: trunk flexion, hip flexion, knee flexion, knee extension, ankle dorsiflexion, and ankle plantar flexion. Surface EMG recordings will be taken from the rectus abdominis, rectus femoris, biceps femoris, vastus lateralis, tibialis anterior, soleus, and gastrocnemius. The root mean square (RMS) EMG amplitude from each muscle during rest and the attempted contraction for each participant and each trial will be calculated to explore presence of muscle activity in each movement.
Change in attempted voluntary motor activation (walking) | Weeks 2 and 14
  Participants will attempt to voluntarily activate lower limb muscles while walking in the body-weight-supported treadmill system. Surface EMG recordings will be taken from the rectus femoris, biceps femoris, vastus lateralis, tibialis anterior, soleus, and gastrocnemius. The root mean square (RMS) EMG amplitude from each muscle during rest and stepping for each participant and each trial will be calculated to explore presence of muscle activity during walking.
Change in lower limb proprioceptive sense | Weeks 2 and 14
  Lower limb proprioceptive sense will be quantified using previously validated assessments of joint position sense and movement detection sense using custom software of the Lokomat. Kinesthesia and joint position sense will be determined.
Change in blood pressure regulation | Weeks 2 and 14
  Blood pressure variability will be measured using a 24-hour ambulatory blood pressure monitor (24-Hr ABPM) which records blood pressure every 15 minutes during the daytime period, and then every hour during the night-time period. Changes in systolic blood pressure will be determined.

SECONDARY OUTCOMES:
Change in corticospinal excitability | Weeks 2 and 14
  Transcranial magnetic stimulation (TMS) will be delivered over the primary motor cortex to elicit motor evoked potentials (MEPs) in the tibialis anterior and soleus muscles. MEPs will be recorded with surface EMG. The amplitude of MEPs will be extracted and plotted against TMS intensity to create a stimulation response curve.
Change in spinal excitability | Weeks 2 and 14
  Motor responses to peripheral nerve stimulation will be measured using surface EMG at the gastrocnemius and soleus muscles. To investigate the changes in spinal reflex excitability, we will examine the size of the H-reflex normalized by M max (H-M ratio) and H-reflex recruitment curves at rest.
Change in seated, static balance control | Weeks 2 and 14
  Balance control will be measured while participants are seated on a force plate with their feet off the floor and arms crossed at their chest. Force plate data will be used to calculate overall seated stability and the amount of postural activity during the task.
Change in seated, dynamic balance control | Weeks 2 and 14
  Balance control will be measured while participants are seated on a force plate with their feet off the floor and arms crossed at their chest. Participants will be asked to lean as far as they can in the 8-cardinal directions. Total distance traveled in each direction as calculated by the center of pressure trajectory from the force plate will be recorded.
Change in severity of cardiovascular dysfunction by the ADFSCI | Weeks 2 and 14
  Autonomic Dysfunction Following Spinal Cord Injury (ADFSCI) questionnaire assesses self-reported frequency and severity of blood pressure dysregulation. The participant will complete 18 items from the third and fourth part of the questionnaire only, which evaluates autonomic dysreflexia and hypotension. A total score will be calculated for each dysfunction.
Change in severity of orthostatic hypotension | Weeks 2 and 14
  Orthostatic hypotension will be measured using a 60-degree head-up tilt table test where the participant's blood pressure will be measured at supine rest for 10 minutes, and then at approximately 60° upright stand position for 15 minutes. Postural changes in systolic blood pressure will be determined.
Change in cardiac structure and function | Weeks 2 and 14
  Cardiac outcomes will be measured using echocardiogram. The echocardiogram images will be collected using parasternal long and short axis, apical 4, 2 and 3 chamber, and subcostal views. Indices will be determined from the mean of three cardiac cycles and will include measures of left ventricular structure, global systolic and diastolic function, and cardiac mechanics.
Change in lower urinary tract function measured by the NBSS | Weeks 2 and 14
  Neurogenic Bladder Symptom Score (NBSS) questionnaire comprises 23 questions covering 3 domains, including incontinence, storage & voiding, and specific consequences, as well as one question on QoL. All scores, for each domain and a total, will be transformed into a continuous scale value.
Change in lower urinary tract function measured by the I-QOL | Weeks 2 and 14
  Incontinence - Quality Of Life (I-QOL) questionnaire comprises 10 questions covering 3 domains, including avoidance and limiting behaviour, psychosocial impacts, and social embarrassment, which will be summarized as a total score.
Change in bowel function measured by the NBDS | Weeks 2 and 14
  Neurogenic Bowel Dysfunction Score (NBDS) questionnaire comprises 10 questions focusing on defecation, constipation, fecal incontinence, and peri-anal skin problems. The consequential NBD score relates to four different neurogenic bowel dysfunction severity levels.
Change in sexual function (for male participants) measured by the IIEF-15 | Weeks 2 and 14
  International Index of Erectile Function (IIEF-15) questionnaire comprises of 15 questions covering five domains, including erectile function, orgasmic function, intercourse satisfaction, and overall satisfaction. Domain scores will be calculated.
Change in sexual function (for female participants) measured by the FSFI | Weeks 2 and 14
  Female Sexual Function Index (FSFI) comprises of 19 questions covering six domains, including desire, arousal, lubrication, orgasm, satisfaction, and pain. Domain and total scores will be calculated.
Change in subjective experience of sexual functioning measured by a semi-structed interview | Weeks 2 and 14
  A sexual health clinician will conduct a semi-structured one-on-one interview to capture the nuances of the subjective experiences of how their sexual functioning has changed over the course of the intervention. Thematic analysis will be conducted using interview transcripts.
Change in fatigue measured by the FSS | Weeks 2 and 14
  Fatigue Severity Scale (FSS) is a 9-item questionnaire, which captures how fatigue interferes with certain activities of daily living and is accompanied by a global fatigue visual analogue scale. A total score will be calculated.
Change in spasticity measured by the SCI-SET | Weeks 2 and 14
  Spinal Cord Injury- Spasticity Evaluation Tool (SCI-SET) is a thorough subjective questionnaire that asks the participant a total of 35 questions regarding both the problematic and useful effects of spasticity on daily life in the past 7 days. A total score will be calculated.
Change in pain measured by the International SCI Pain Basic Data Set (version 2) | Weeks 2 and 14
  The International SCI Pain Basic Data Set Version 2 determines the intensity and location of pain, and the subsequent impact of that pain interference on different domains of life. A total score will be calculated for each domain.
Change in quality of life measured by the SF-36 | Weeks 2 and 14
  Short Form (SF-36) health survey consists of 8 domains pertaining to the participants' experiences in the last 4 weeks, with 4 representing physical quality of life (Physical Component Summary) and 4 representing emotional quality of life (Mental Component Summary) Each of the 8 summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD,PhD,FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Blusson Spinal Cord Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Shackleton C, Samejima S, Williams AM, Malik RN, Balthazaar SJ, Alrashidi A, Sachdeva R, Elliott SL, Nightingale TE, Berger MJ, Lam T, Krassioukov AV. Motor and autonomic concomitant health improvements with neuromodulation and exercise (MACHINE) training: a randomised controlled trial in individuals with spinal cord injury. BMJ Open. 2023 Jul 14;13(7):e070544. doi: 10.1136/bmjopen-2022-070544. PMID 37451734